CLINICAL TRIAL: NCT04015011
Title: A Pilot Study Investigating the Effects of a Three-Month Low Calorie Diet Weight Loss Intervention on Knee Replacement Outcomes
Brief Title: Effects of a Three-Month Low Calorie Diet Weight Loss Intervention on Knee Replacement Outcomes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study enrollment ended early due to covid and lack of continued funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-00319
Record Dates: First submitted 2019-06-26; First posted 2019-07-10 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Calorie Diet (LCD) diet intervention (Experimental): In person or video conference
  Interventions: Combination Product: LCD Intervention

INTERVENTIONS:
Combination Product: LCD Intervention — composed of approximately 1,080 kcal/day, which includes 3 New Direction Meal Replacements containing 200 kcal (27g protein, 12g carbhydrate, 2g fiber), 1 protein bar containing 160 kcal (5 g protein, 18g carbohydrate, 5g fiber, 2g sugar alcohol), and a 350-calorie controlled meal of protein and vegetables that the patient will make on his/ her own.

SUMMARY:
Total Knee Replacement (TKR) significantly improves function, pain, and overall quality of life in patients with end-stage arthritis of the knee. However, studies show that obesity increases complications and costs associated with TKR. The American Academy of Orthopaedic Surgeons (AAOS) clinical guidelines recommend that patients with a BMI > 25kg/m2 lose 5% of their body weight prior to surgery. Consequently, although it is not clear how to patients or providers achieve weight loss in this population, some providers and hospitals decline to perform TKR in patients with obesity. Low Calorie meal replacement diets (LCD) are a feasible way to safely promote short-term weight loss of 8-15% at 3-6 months prior to some elective surgeries.

This is a pilot efficacy study to test whether a short-term program using a 3-month LCD leads to weight loss and improved patient reported and functional outcomes. 75 patients eligible for knee replacement surgery and willing to undergo non-operative weight management treatment at NYU Langone Comprehensive Obesity Center. This study will establish feasibility and weight loss outcomes in preparation for a multicenter effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

* BMI 35-45 kg/m2
* Any ethnicity
* Able to speak, read, and write in English
* Have knee replacement surgery already planned by the surgeon
* Plan to undergo knee replacement surgery within 3-6 months post LCD intervention
* Willing to commute to NYU Langone Weight Management Clinic at the start of the dietary intervention, midway through, and end of intervention

Exclusion Criteria:

* Uncontrolled type 2 diabetes, defined as HbA1c > 9%
* If smokes cigarettes, must go through a 6 week cessation program first
* Type 1 diabetes
* Whey protein allergies
* Soy allergies
* Anyone in whom rapid weight loss is not indicated (e.g., ESRD or cirrhosis, metabolic cancer, abnormal 3 times UL liver enzyme labs)
* Current untreated or uncontrolled eating disorder (e.g., binge eating, bulimia)
* Rheumatoid arthritis
* In case a previous knee replacement surgery was done, the participant should wait at least 1 year from previous date of surgery
* Undergoing simultaneous bilateral knee replacement
* Enrolled in a formal weight loss program
* Taking anti-obesity medications
* Coexisting psychotic conditions requiring hospitalization or more intense treatment (e.g., bipolar mood disorder, severe depression)
* Abnormal CBC, and uric acid, must be treated prior to start of intervention
* Higher than 5.5 mU/L or lower than 0.3 mU/L TSH must be treated prior to start of LCD intervention

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in weight | up to 18 Months
  Patients who have had recent knee replacement will be weighed at screening, week 5-7, week 11-13, and 30-120 days post surgery
Change in mobility during 30-sec chair stand | 18 Months
Change in mobility during 40-meter fast paced walk | 18 Months
Change in quality of life measured by SF-36 questionnaire | 18 Months
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software. Pricing depends on the number of scores that the researcher needs to calculate.
  The eight sections are:
  * vitality
  * physical functioning
  * bodily pain
  * general health perceptions
  * physical role functioning
  * emotional role functioning
  * social role functioning
  * mental health

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Langone Health, New York, New York, United States